CLINICAL TRIAL: NCT00603369
Title: HIV, Abuse, and Psychiatric Disorders Among Youth
Acronym: Project STAR
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Rhode Island Hospital (Other)
Responsible Party: Larry K. Brown/Principal Investigator, Rhode Island Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R01MH061149 (NIH); R01MH061149 (NIH)
Record Dates: First submitted 2008-01-16; First posted 2008-01-29 (Estimated); Last update posted 2009-02-06 (Estimated); Status verified 2009-02

CONDITIONS: HIV Infections
Keywords: HIV prevention; HIV seronegativity
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): 13 session group intervention including sexual health information, affect management skills, cognitive monitoring, and communication skills training.
  Interventions: Behavioral: group intervention
- 2 (Active Comparator): 2 session group intervention including sexual health information training.
  Interventions: Behavioral: group intervention

INTERVENTIONS:
Behavioral: group intervention — 13-session intervention
  Arms: 1
Behavioral: group intervention — 2-session intervention
  Arms: 2

SUMMARY:
One subgroup of adolescents at particular risk for HIV is those with psychiatric disorders. Furthermore, those with histories of sexual abuse have been found to have riskier attitudes, poorer sexual communication skills, and less consistent condom use than non-abused peers. This study implemented and evaluated interventions for adolescents in intensive psychiatric treatment settings, particularly those with histories of sexual abuse. It is hypothesized that those participating in the intervention that addresses affect management and cognitive monitoring strategies will show fewer HIV-risk related behaviors and attitudes at posttest than peers in an information-based intervention.

ELIGIBILITY:
Inclusion Criteria:

* Adolescent attending therapeutic school

Exclusion Criteria:

* Adolescent is HIV positive
* Adolescent is developmentally delayed
* Adolescent is pregnant
* Adolescent has a history of sexual crime

Ages: 13 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 212 (Actual)
Dates: Start 1999-09; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
condom use | 1 year

SECONDARY OUTCOMES:
scores on HIV knowledge questionnaire | 1 year
number of sexual partners | 1 year
scores on measure of attitudes toward condom use | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Larry K. Brown, MD, Principal Investigator — Rhode Island Hospital
Locations (1):
- Rhode Island Hospital, Providence, Rhode Island, United States

REFERENCES:
- [Derived] Brown LK, Nugent NR, Houck CD, Lescano CM, Whiteley LB, Barker D, Viau L, Zlotnick C. Safe Thinking and Affect Regulation (STAR): human immunodeficiency virus prevention in alternative/therapeutic schools. J Am Acad Child Adolesc Psychiatry. 2011 Oct;50(10):1065-74. doi: 10.1016/j.jaac.2011.06.018. Epub 2011 Aug 27. PMID 21961780